CLINICAL TRIAL: NCT05204784
Title: A Randomized Controlled Prospective Single-center Feasibility Study of Rheopheresis for Raynaud's Syndrome and Digital Ulcers in Systemic Sclerosis
Brief Title: Rheopheresis for Raynaud's and Digital Ulcers in Systemic Sclerosis
Acronym: RHEACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter Korsten (Other)
Collaborators: DiaMed GmbH (Industry)
Responsible Party: Sponsor-Investigator, Peter Korsten, Dr. med., University of Göttingen
Organization: University of Göttingen (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 36/7/21
Record Dates: First submitted 2021-11-29; First posted 2022-01-24 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Systemic Sclerosis; Raynaud Phenomenon; Digital Ulcer; Scleroderma
Keywords: Rheopheresis; Raynaud Phenomenon; Systemic Sclerosis; Digital Ulcers; Therapeutic plasma exchange
MeSH Terms: conditions — Scleroderma, Systemic; Raynaud Disease; digital ulcers; Scleroderma, Diffuse | interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): 2 Rheopheresis treatments per week x 2, followed by 8 weeks without treatment, 8 overall treatments
  Interventions: Procedure: Rheopheresis treatment
- Arm 2 (Experimental): 2 Rheopheresis treatments in week 1, followed by 1 treatment every 2 weeks, 8 overall treatments
  Interventions: Procedure: Rheopheresis treatment
- Control Group (Active Comparator): Standard of care treatment with intravenous iloprost
  Interventions: Drug: Intravenous Infusion

INTERVENTIONS:
Procedure: Rheopheresis treatment — After obtaining venous access, anticoagulated blood is pumped through a plasmafilter. The plasma is then run through the Rheofilter and large plasma proteins are removed. Finally, cells are reinfused, and blood is returned to the patient.
  Arms: Arm 1; Arm 2
Drug: Intravenous Infusion — Standard of care treatment consists of intravenous iloprost infusions at a dose of 0.5-2 ng/kg/min administered over at least 6 hours as per local standard
  Arms: Control Group

SUMMARY:
In this feasibility study, we aim to explore therapeutic Rheopheresis (RheoP) as a novel treatment option for SSc-associated Raynaud's phenomenon and/or digital ulcers and compare it to the standard of care treatment (intravenous iloprost. RheoP has been used for RP/DU with some success in observational studies, nevertheless, the optimal treatment modality, duration, or frequency of RheoP (and PEX in general) in SSc has not been established as of yet.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients fulfilling ACR/EULAR classification criteria for SSc
2. Presence of RP with or without DU
3. Failure of at least one standard of care treatment (CCB or iloprost) for at least three months
4. RCS > 4
5. Possibility to obtain venous access (either through a peripherally or centrally inserted catheter)

Exclusion Criteria:

1. Significant anemia (<8 g/dL)
2. Clinically relevant hemorrhagic diathesis or coagulopathy
3. Diabetes mellitus
4. Serious acute or chronic kidney (eGFR<30 ml/min/1.73m2) or liver failure
5. Hypotension with systolic blood pressure <100 mmHg
6. Chronic viral infections (HIV, Hepatitis B, C)
7. Epilepsia, psychosis, dementia, or other relevant neurologic condition precluding the conduct of plasmapheresis
8. Malignant disease or any other condition with life expectancy <12 months
9. Known history of alcohol or drug abuse
10. Long-term serious tobacco abuse with documented severe vascular disease (Fontaine >III).
11. Severe hyperlipoproteinemia, defined as a significant elevation of Lp(a) or LDL cholesterol despite standard doses of medical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Raynaud Condition Score (RCS) | 24 weeks
  changes of the Raynaud Condition after treatment, higher RCS denotes worse clinical findings

SECONDARY OUTCOMES:
Development of new digital ulcers | 24 weeks
  To assess the number of new digital ulcers with treatment
Time to healing of existing digital ulcers | 24 weeks
  Time to healing of existing digital ulcers
Scleroderma Health Assessment Questionnaire | 24 weeks
  Changes in the SHAQ with treatment; higher scores mean better functional status
Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue score | 24 weeks
  changes in the FACIT-Fatigue score with treatment; higher scores indicate a better clinical status
Quick DASH | 24 weeks
  changes in the Quick DASH with treatment; lower scores mean better functional status
Nailfold video capillaroscopy changes | 24 weeks
  changes in in NVC assessments with treatment
Whole blood viscosity | 24 weeks
  changes in Whole blood viscosity with treatment

OTHER OUTCOMES:
Exploratory objectives | 24 weeks
  changes in miRNA

CONTACTS AND LOCATIONS:
Overall Officials: Peter Korsten, Dr. med., Principal Investigator — University Medical Center Göttingen
Locations (1):
- University Medical Center Göttingen, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wigley FM. Clinical practice. Raynaud's Phenomenon. N Engl J Med. 2002 Sep 26;347(13):1001-8. doi: 10.1056/NEJMcp013013. No abstract available. PMID 12324557
- [Background] Gabrielli A, Avvedimento EV, Krieg T. Scleroderma. N Engl J Med. 2009 May 7;360(19):1989-2003. doi: 10.1056/NEJMra0806188. No abstract available. PMID 19420368
- [Background] Allanore Y, Simms R, Distler O, Trojanowska M, Pope J, Denton CP, Varga J. Systemic sclerosis. Nat Rev Dis Primers. 2015 Apr 23;1:15002. doi: 10.1038/nrdp.2015.2. PMID 27189141
- [Background] Abraham S, Steen V. Optimal management of digital ulcers in systemic sclerosis. Ther Clin Risk Manag. 2015 Jun 15;11:939-47. doi: 10.2147/TCRM.S82561. eCollection 2015. PMID 26109864
- [Background] Herrick AL. Management of Raynaud's phenomenon and digital ischemia. Curr Rheumatol Rep. 2013 Jan;15(1):303. doi: 10.1007/s11926-012-0303-1. PMID 23292819
- [Background] Matucci-Cerinic M, Denton CP, Furst DE, Mayes MD, Hsu VM, Carpentier P, Wigley FM, Black CM, Fessler BJ, Merkel PA, Pope JE, Sweiss NJ, Doyle MK, Hellmich B, Medsger TA Jr, Morganti A, Kramer F, Korn JH, Seibold JR. Bosentan treatment of digital ulcers related to systemic sclerosis: results from the RAPIDS-2 randomised, double-blind, placebo-controlled trial. Ann Rheum Dis. 2011 Jan;70(1):32-8. doi: 10.1136/ard.2010.130658. Epub 2010 Aug 30. PMID 20805294
- [Background] Korsten P, Niewold TB, Zeisberg M, Utset TO, Cho D, Zachary LS, Sweiss NJ, Volkov S. Increased Whole Blood Viscosity Is Associated with the Presence of Digital Ulcers in Systemic Sclerosis: Results from a Cross-Sectional Pilot Study. Autoimmune Dis. 2017;2017:3529214. doi: 10.1155/2017/3529214. Epub 2017 Nov 29. PMID 29318042
- [Background] Koss MJ, Kurz P, Tsobanelis T, Lehmacher W, Fassbender C, Klingel R, Koch FH. Prospective, randomized, controlled clinical study evaluating the efficacy of Rheopheresis for dry age-related macular degeneration. Dry AMD treatment with Rheopheresis Trial-ART. Graefes Arch Clin Exp Ophthalmol. 2009 Oct;247(10):1297-306. doi: 10.1007/s00417-009-1113-7. Epub 2009 Jul 23. PMID 19629514
- [Background] Kostal M, Drsata J, Blaha M, Lanska M, Chrobok V. Rheopheresis in treatment of idiopathic sensorineural sudden hearing loss. J Otolaryngol Head Neck Surg. 2017 Jun 29;46(1):50. doi: 10.1186/s40463-017-0228-9. PMID 28662721
- [Background] Klingel R, Erdtracht B, Gauss V, Piazolo A, Mausfeld-Lafdhiya P, Diehm C. Rheopheresis in patients with critical limb ischemia--results of an open label prospective pilot trial. Ther Apher Dial. 2005 Dec;9(6):473-81. doi: 10.1111/j.1744-9987.2005.00276.x. PMID 16354279
- [Background] Klingel R, Mumme C, Fassbender T, Himmelsbach F, Altes U, Lotz J, Pohlmann T, Beyer J, Kustner E. Rheopheresis in patients with ischemic diabetic foot syndrome: results of an open label prospective pilot trial. Ther Apher Dial. 2003 Aug;7(4):444-55. doi: 10.1046/j.1526-0968.2003.00082.x. PMID 12887730
- [Background] Harris ES, Meiselman HJ, Moriarty PM, Metzger A, Malkovsky M. Therapeutic plasma exchange for the treatment of systemic sclerosis: A comprehensive review and analysis. J Scleroderma Relat Disord. 2018 Jun;3(2):132-152. doi: 10.1177/2397198318758606. Epub 2018 Mar 9. PMID 35382237
- [Background] Schwartz J, Padmanabhan A, Aqui N, Balogun RA, Connelly-Smith L, Delaney M, Dunbar NM, Witt V, Wu Y, Shaz BH. Guidelines on the Use of Therapeutic Apheresis in Clinical Practice-Evidence-Based Approach from the Writing Committee of the American Society for Apheresis: The Seventh Special Issue. J Clin Apher. 2016 Jun;31(3):149-62. doi: 10.1002/jca.21470. PMID 27322218
- [Background] Khanna D, Lovell DJ, Giannini E, Clements PJ, Merkel PA, Seibold JR, Matucci-Cerinic M, Denton CP, Mayes MD, Steen VD, Varga J, Furst DE; Scleroderma Clinical Trials Consortium co-authors. Development of a provisional core set of response measures for clinical trials of systemic sclerosis. Ann Rheum Dis. 2008 May;67(5):703-9. doi: 10.1136/ard.2007.078923. Epub 2007 Sep 24. PMID 17893248
- [Background] Cutolo M, Smith V, Furst DE, Khanna D, Herrick AL. Points to consider-Raynaud's phenomenon in systemic sclerosis. Rheumatology (Oxford). 2017 Sep 1;56(suppl_5):v45-v48. doi: 10.1093/rheumatology/kex199. PMID 28992170
- [Background] Wigley FM, Wise RA, Seibold JR, McCloskey DA, Kujala G, Medsger TA Jr, Steen VD, Varga J, Jimenez S, Mayes M, Clements PJ, Weiner SR, Porter J, Ellman M, Wise C, Kaufman LD, Williams J, Dole W. Intravenous iloprost infusion in patients with Raynaud phenomenon secondary to systemic sclerosis. A multicenter, placebo-controlled, double-blind study. Ann Intern Med. 1994 Feb 1;120(3):199-206. doi: 10.7326/0003-4819-120-3-199402010-00004. PMID 7506013
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Ellen Csuka M, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American college of rheumatology/European league against rheumatism collaborative initiative. Ann Rheum Dis. 2013 Nov;72(11):1747-55. doi: 10.1136/annrheumdis-2013-204424. PMID 24092682
- [Background] Merkel PA, Herlyn K, Martin RW, Anderson JJ, Mayes MD, Bell P, Korn JH, Simms RW, Csuka ME, Medsger TA Jr, Rothfield NF, Ellman MH, Collier DH, Weinstein A, Furst DE, Jimenez SA, White B, Seibold JR, Wigley FM; Scleroderma Clinical Trials Consortium. Measuring disease activity and functional status in patients with scleroderma and Raynaud's phenomenon. Arthritis Rheum. 2002 Sep;46(9):2410-20. doi: 10.1002/art.10486. PMID 12355489
- [Derived] Rademacher JG, Tampe B, Borisch A, Buschfort RM, von Figura A, Asendorf T, Korsten P. Study Protocol: A Randomized Controlled Prospective Single-Center Feasibility Study of Rheopheresis for Raynaud's Syndrome and Digital Ulcers in Systemic Sclerosis (RHEACT Study). Front Med (Lausanne). 2022 Apr 14;9:871744. doi: 10.3389/fmed.2022.871744. eCollection 2022. PMID 35492333